CLINICAL TRIAL: NCT04438512
Title: An Intermediate-size Multi-site Expanded Access Program for MDMA-assisted Psychotherapy for Patients With Treatment-resistant PTSD
Brief Title: A Multi-site Expanded Access Program for MDMA-assisted Psychotherapy for Patients With Treatment-resistant PTSD
Acronym: EAMP1
Status: No longer available | Type: Expanded Access
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: EA
Record Dates: First submitted 2020-02-25; First posted 2020-06-18 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Midomafetamine — Administration of 80 or 120 mg midomafetamine HCl in combination with manualized therapy and a supplemental dose 1.5 to 2 hrs later of 40 or 60 mg midomafetamine HCl, respectively
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine HCl
Behavioral: Psychotherapy — Manualized therapy performed by therapist team

SUMMARY:
The goal of this expanded access protocol is to provide access to MDMA-assisted therapy for eligible patients with treatment-resistant PTSD who are not able to enroll in another MDMA-assisted therapy clinical trial.

Participants will undergo three non-drug preparatory therapy sessions followed by three MDMA-assisted therapy sessions. Each MDMA-assisted therapy session will be followed by three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This is an open-label, expanded access protocol for eligible patients with treatment-resistant PTSD. This protocol is designed to provide access to MDMA-assisted therapy for patients who are not eligible for participation in another ongoing MDMA-assisted therapy clinical trial. In addition, this program will provide supportive data on safety and tolerability of MDMA-assisted therapy in treatment-resistant patients with PTSD. The study will treat up to 50 patients.

A flexible dose of MDMA (80 to 120 mg midomafetamine HCl), followed by a supplemental dose unless contraindicated, is administered during the Treatment Period with manualized therapy in up to three open-label Experimental Sessions. During the Treatment Period, each Experimental Session is preceded by three 90-minute Preparatory Sessions and followed by three 90-minute Integrative Sessions of non-drug therapy. Experimental Sessions will be followed by an overnight stay.

ELIGIBILITY:
Inclusion Criteria:

* At Screening, meet criteria for PTSD diagnosis according to medical history and clinical interview and have at least moderate PTSD symptoms in the last month.
* Have had at least two unsuccessful attempts at treatment for PTSD. Treatment attempts can consist of adequate dose and duration of medication treatment (at least 3 months of Paroxetine or Sertraline or other SSRI at dosages recommended in the package insert) or adequate duration of therapy treatment (at least 12 sessions of psychotherapy) or any combination of these two categories.
* Are at least 18 years old.
* Are fluent in speaking and reading a recognized language of the expanded access site.
* Are able to swallow pills.
* Agree to have study visits recorded, if applicable, including Experimental Sessions and non-drug therapy sessions.
* Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a patient becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If a patient has the ability to become pregnant, they must have a negative pregnancy test at program entry and prior to each Experimental Session, and must agree to use adequate contraception through 10 days after the last Experimental Session.
* Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not participate in any other interventional clinical trials during the duration of the protocol without prior approval of the medical monitor, remain overnight at the site, or nearby location, after each Experimental Session and be driven home on the following day, and commit to medication dosing, therapy, and program procedures.
* May have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines, if they pass additional screening within the past year to rule out underlying cardiovascular disease.
* May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
* May have current alcohol or substance use disorder if patient meets criteria for early remission prior to enrollment.
* May have a history of or current Diabetes Mellitus (Type 1 or Type 2), if the patient passes additional screening to rule out underlying cardiovascular disease
* May have hypothyroidism if taking adequate and stable thyroid replacement medication.
* May have a history of, or current glaucoma, if approval for program participation is received from an ophthalmologist.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have any current problem which, in the opinion of the investigator or medical monitor, might interfere with participation.
* Have used Ecstasy (material represented as containing MDMA) within three months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial.
* In the investigator's opinion, lack a stable living situation or supportive family/network.
* Have evidence or history of significant medical and psychiatric disorders.
* Any patient presenting current serious suicide risk.
* Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist.
* Have evidence or history of significant hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of MDMA.
* Have a history of ventricular arrhythmia, other than occasional PVCs in the absence of ischemic heart disease, at any time or with a history of supraventricular arrhythmia within the past year.
* Have a diagnosis of uncontrolled hypertension using the standard criteria of the American Heart Association for Stage 2 hypertension (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions).
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males or >460 ms in females corrected by Fridericia's formula).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions.
* Have symptomatic liver disease or have significant liver enzyme elevation.
* Have a history of HCV that has not been evaluated and treated successfully if treatment is indicated.
* Have history of hyponatremia or hyperthermia.
* Are pregnant or nursing, or able to become pregnant and are not practicing an effective means of contraception.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Manish Agrawal, MD, Principal Investigator — Sunstone Medical, PC; Caroline Lewis, MD, Principal Investigator — Pearl Psychedelic Institute
Locations (2):
- United States (2):
  - Sunstone Medical, PC, Rockville, Maryland
  - Pearl Psychedelic Institute, Waynesville, North Carolina